CLINICAL TRIAL: NCT02012777
Title: Propanolol Effect on Red Cell Adhesion in Non-Asthmatic Children With Sickle Cell Disease: A Dose Finding Study
Brief Title: Propanolol and Red Cell Adhesion Non-asthmatic Children Sickle Cell Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to recruit patients into the study.
Sponsor: University of Miami (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Ofelia Alvarez, Professor of Clinical Pediatrics, University of Miami
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100334
Record Dates: First submitted 2013-12-06; First posted 2013-12-16 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; propanolol; red blood cell adhesion
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Propranolol; propranolol CR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cohort 1 10mg propranolol (Active Comparator): first study arm will consist of 5 subjects who will be administered a dose of 10mg propanolol and followed 1-4 weeks.
  Data safety and monitoring committee has reviewed the data for safety and instructed the study to continue based on the findings.
  Interventions: Drug: propranolol
- cohort 2 20mg propranolol (Active Comparator): This cohort will involve the administration of 5 subjects with 20mg propanolol. The data safety and monitoring committee will review the data for safety when the 5 subjects are recruited and instruct the study to continue depending on the findings.
  Interventions: Drug: propranolol
- cohort 3 40mg propranolol (Active Comparator): This cohort will involve the administration of 10 subjects with 40mg propanolol. The data safety and monitoring committee will review the data for safety when the 10 subjects are recruited and instruct the study to continue depending on the findings.
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: propranolol — Propranolol hydrochloride is a synthetic beta-adrenergic receptor-blocking agent. This will be administered in an open-label single administration to 3 cohorts (10mg, 20mg, and 40mg) of children with sickle cell disease. Patient blood will be evaluated for red cell adhesion and patient data evaluated for safety monitoring.
  Other Names: propanolol systemic; Inderal; Inderal LA; InnoPran XL

SUMMARY:
Propanolol is a beta blocker which has been found to inhibit the ability of epinephrine to upregulate sickle red cell adhesion to laminin and endothelial cells in vitro. The purpose of this pilot study is to administer one dose of propanolol to children with sickle cell disease and to measure pre and post dose red cell adhesion. The hypothesis is that a single dose of propanolol will decrease red cell adhesion to laminin and endothelial cells as compared to baseline.

DETAILED DESCRIPTION:
A similar pilot study has already been conducted in adults and is now being tried in children to gather preliminary data for a grant submission. No safety issues were found in the adult pilot study. This study will evaluate the effect of different doses of propanolol. The risks of this study involve the risks of three (3) blood draws and the risks of propanolol. In order to minimize the risks children with sickle cell disease and asthma will be excluded because asthma is a contraindication to the use of propanolol. In addition, patients will not be hypertensive or bradycardic.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of HbSS or HbSBeta0Thal
2. age 10-17 years
3. Weight 30kg or greater
4. Hb 7mg/dL or greater
5. informed consent

Exclusion Criteria:

1. History of vaso-occlusive crisis during the past 6 weeks, or history of transfusion during the past 3 months.
2. pregnancy
3. history of heart failure, myocardial infarction, asthma, bradyarrythmias, hypotension, thyroid disease, diabetes, renal insufficiency
4. concurrent medications: any antihypertensive medication, diuretics, thyroid replacement medications, any arrythmia medication, insulin, hypoglycaemic medication
5. history of allergy to sulfonamides
6. elevated BUN or creatinine

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2013-04-03 (Actual)

PRIMARY OUTCOMES:
measurement of the sickle red cell response to epinephrine | 1-4 weeks
  At study initiation 5mL of blood is drawn to evaluate for red cell adhesion (screening visit or visit 1). At the intervention visit 1-4 weeks later another 5mL of blood will be drawn and patient will have an ECG performed, followed by one dose of propanolol at the stratum that s/he is in. Vitals signs will be monitored (including blood pressure) for 4 hours after drug administration.

SECONDARY OUTCOMES:
Safety data regarding the use of propanolol in children with sickle cell disease | within 24 hours after drug administration
  1. New onset wheezing
  2. Onset of low blood pressure defined as blood pressure less than 90/50
  3. Onset of heart rate less than 60 beats/min

CONTACTS AND LOCATIONS:
Overall Officials: Ofelia A Alvarez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Storch CH, Hoeger PH. Propranolol for infantile haemangiomas: insights into the molecular mechanisms of action. Br J Dermatol. 2010 Aug;163(2):269-74. doi: 10.1111/j.1365-2133.2010.09848.x. Epub 2010 May 8. PMID 20456345
- [Result] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Result] Lawley LP, Siegfried E, Todd JL. Propranolol treatment for hemangioma of infancy: risks and recommendations. Pediatr Dermatol. 2009 Sep-Oct;26(5):610-4. doi: 10.1111/j.1525-1470.2009.00975.x. PMID 19840322
- [Result] Zimmermann AP, Wiegand S, Werner JA, Eivazi B. Propranolol therapy for infantile haemangiomas: review of the literature. Int J Pediatr Otorhinolaryngol. 2010 Apr;74(4):338-42. doi: 10.1016/j.ijporl.2010.01.001. Epub 2010 Feb 1. PMID 20117846
- [Result] Lamy S, Lachambre MP, Lord-Dufour S, Beliveau R. Propranolol suppresses angiogenesis in vitro: inhibition of proliferation, migration, and differentiation of endothelial cells. Vascul Pharmacol. 2010 Nov-Dec;53(5-6):200-8. doi: 10.1016/j.vph.2010.08.002. Epub 2010 Aug 20. PMID 20732454
- [Result] Holmes WJ, Mishra A, Gorst C, Liew SH. Propranolol as first-line treatment for rapidly proliferating infantile haemangiomas. J Plast Reconstr Aesthet Surg. 2011 Apr;64(4):445-51. doi: 10.1016/j.bjps.2010.07.009. Epub 2010 Aug 24. PMID 20797926
- [Result] Schiestl C, Neuhaus K, Zoller S, Subotic U, Forster-Kuebler I, Michels R, Balmer C, Weibel L. Efficacy and safety of propranolol as first-line treatment for infantile hemangiomas. Eur J Pediatr. 2011 Apr;170(4):493-501. doi: 10.1007/s00431-010-1324-2. Epub 2010 Oct 9. PMID 20936416
- [Result] Chang, MW. Journal Watch Dermatology. Nov 6, 2009 Propanolol for Infantile Hemangioma: Safety Issues and Proposed Protocol
- [Result] Holland KE, Frieden IJ, Frommelt PC, Mancini AJ, Wyatt D, Drolet BA. Hypoglycemia in children taking propranolol for the treatment of infantile hemangioma. Arch Dermatol. 2010 Jul;146(7):775-8. doi: 10.1001/archdermatol.2010.158. PMID 20644039